CLINICAL TRIAL: NCT02524301
Title: Evaluation of Brain Opioid Receptor Activity in Anorexia Nervosa : a PET [11C]Diprenorphine Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0908019
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Body Dysmorphic Disorders; Anorexia
Keywords: anorexia nervosa; opioid receptors; Positron emission tomography (PET); diprenorphine
MeSH Terms: conditions — Body Dysmorphic Disorders; Anorexia; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anorexia nervosa patients (Experimental): Cerebral [11C]diprenorphine Binding Potential measured by Positron emission Tomography (PET)
  Interventions: Drug: Positron Emission Tomography using [11C]diprenorphine
- Recovered anorexia nervosa patients (Experimental): Cerebral [11C]diprenorphine Binding Potential measured by Positron emission Tomography (PET)
  Interventions: Drug: Positron Emission Tomography using [11C]diprenorphine
- Healthy Volonteers (Experimental): Cerebral [11C]diprenorphine Binding Potential measured by Positron emission Tomography (PET)
  Interventions: Drug: Positron Emission Tomography using [11C]diprenorphine

INTERVENTIONS:
Drug: Positron Emission Tomography using [11C]diprenorphine — PET using [11C]diprenorphine
  Other Names: PET

SUMMARY:
The place of opioid system in anorexia nervosa (AN) physiopathology is still unclear. Conflicting results were published on cerebral spinal fluid or peripheral levels in anorexia nervosa. However, no data have been reported on opioid cerebral activity. Diprenorphine is a ligand with non-selective binding to opiate receptors µ, κ and δ capable to assess the interaction between endogenous opioids and their receptors.

ELIGIBILITY:
Inclusion Criteria:

* AN patients DSM IV criteria including amenorrhea BMI < 17.5 kg/m² and abnormal nutritional markers Group 1 (N=15) : long period of / recurrent weight loss (> 2 yrs) Group 2 (N=15) : recent weight loss (6 to 12 months)
* Recovered AN patients History of AN Weight recovery and BMI > 18.5 kg/m², stable for at least 12 months Normal nutritional markers Group 1 (N=15) : menses recovery after bodyweight stabilization Group 2 (N=15) : long persistence of amenorrhea (> 12 months) despite weight recovery
* Healthy volunteers (N=15) BMI between 18.5 and 25 kg/m², normal nutritional markers, absence of psychiatric or organic pathology
* For all subjects Women 18-35 yrs Written and sign consent Affiliation to health insurance

Exclusion Criteria:

* History of heart failure
* Psychotropic treatment , antiepileptics
* Ongoing or suspected pregnancy, positive beta HCG test before brain imaging
* Intense physical activity
* Constrains for MRI (ferromagnetic implants or claustrophobia)
* Refusal to be informed in case of incidentaloma revealed by brain imaging
* Refusal for written consent

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
[11C]diprenorphine binding potential | week 2
  Value of [11C]diprenorphine binding potential (BP) in predefined brains regions [11C] diprenorphine BP will be evaluated by brain positron emission tomography

SECONDARY OUTCOMES:
Correlation [11C]diprenorphine binding potential | week 2
  Correlation between [11C]diprenorphine binding potential and plasma endogenous opioid levels
Correlation [11C]diprenorphine binding potential | week 2
  Correlation between [11C]diprenorphine binding potential and psychometric score evaluating addictive behavior, reward and positive reinforcement
Correlation [11C]diprenorphine binding potential | week 2
  Correlation between [11C]diprenorphine binding potential and appetite regulating hormones
Correlation [11C]diprenorphine binding potential | week 2
  Correlation between [11C]diprenorphine binding potential and LH response during GnRH test

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Estour, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (3):
- France (3):
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CNRH, Clermont-Ferrand
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galusca B, Traverse B, Costes N, Massoubre C, Le Bars D, Estour B, Germain N, Redoute J. Decreased cerebral opioid receptors availability related to hormonal and psychometric profile in restrictive-type anorexia nervosa. Psychoneuroendocrinology. 2020 Aug;118:104711. doi: 10.1016/j.psyneuen.2020.104711. Epub 2020 May 19. PMID 32460196